CLINICAL TRIAL: NCT01534039
Title: Phase 4-A Clinical Comparison of a Marketed Moldable Skin Barrier Versus a Marketed Stretch-to-Fit Skin Barrier in Healthy Volunteers
Brief Title: A Clinical Comparison of Two Marketed Skin Barriers on Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Independent Nurse Consultants LLC (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: INC#001
Record Dates: First submitted 2011-12-19; First posted 2012-02-16 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Peristomal Skin Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sur-Fit Natura/FormaFlex (Active Comparator): Subject will be on Surfit Moldable for 2 weeks then crossover to Formaflex
  Interventions: Device: Sur-Fit Natura
- FormaFlex/Sur-Fit Natura (Active Comparator): Subject will be on Formaflex for 2 weeks then crossover to Surfit Moldable
  Interventions: Device: FormaFlex

INTERVENTIONS:
Device: Sur-Fit Natura — ConvaTec Moldable Skin Barrier for ostomy patients
  Other Names: ConvaTec Moldable Skin Barrier
  Arms: Sur-Fit Natura/FormaFlex
Device: FormaFlex — Hollister skin barrier for ostomy patients
  Other Names: Hollister FormaFlex
  Arms: FormaFlex/Sur-Fit Natura

SUMMARY:
A comparison of two skin barriers on healthy volunteers with a colostomy, ileostomy or urostomy.

Endpoints of comparison include the ability to maintain a secure fit around the stoma, skin protection, wear-time, ease of use, ease of teaching, and comfort.

DETAILED DESCRIPTION:
Study to include 60 subjects, three centers, total of 4 weeks, 2 weeks in each product. Subjects recruited from a population of persons who have had an existing fecal or urinary stoma for a duration of at least three months. There is no restriction on primary diagnosis for ostomy surgery. Subjects must be of legal consenting age, must currently be managing their own stoma with a two piece pouching system, either a pre-cut, cut to fit, moldable or stretch-to-fit, any manufacturer. Subjects may not require convexity and be willing to not to use any accessory products during the study.

ELIGIBILITY:
Inclusion Criteria:

* Existing fecal or urinary ostomy for at least three months,consenting age, able to perform independent ostomy care, willing to not use accessory products, currently wearing a 2 piece marketed product.
* Able to participate for four weeks.

Exclusion Criteria:

* Needing convexity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Ability to maintain secure (snug) fit around stoma | Two weeks
  1. Subject assessment of barrier fit based on questionnaire at each skin barrier change up to 2 weeks
  2. Barrier gap assessment performed by nurse at 2 weeks
  3. Barrier gap assessment performed by subject at each skin barrier change up to 2 weeks

SECONDARY OUTCOMES:
Skin Protection | Two weeks
  1. SACS assessment by patient at each barrier change up to 2 weeks
  2. SACS assessment by nurse at 2 weeks
Wear Time | Two weeks
  1. Time of barrier change recorded
Ease of use | Two weeks
  1. Assessment by subject response to questionnaire
Ease of teaching | Two weeks
  1. Assessment by nurse of ability to teach subject to use barrier
Comfort | Two weeks
  1. Subject assessment of comfort of barrier at each change

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Durnal, RN BSN WOCN, Principal Investigator — Independent Nurse Consultants LLC
Locations (1):
- Independent Nurse Consultants LLC, Tucson, Arizona, United States